CLINICAL TRIAL: NCT06900244
Title: Probing Metabolic Dysregulation and Altered Substrate Metabolism in the Healthy and Disrupted Brain Using Hyperpolarised 13C Labelled Substrates.
Brief Title: Metabolic Imaging of Neurological Disease
Acronym: MIND
Status: Enrolling by invitation | Type: Observational
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Other Study IDs: 281106
Record Dates: First submitted 2025-03-17; First posted 2025-03-28 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Multiple Sclerosis: All phenotypes

SUMMARY:
Multiple Sclerosis is a chronic condition that shows changes in the way that the brain consumes sugar. It is also known that there are a number of metabolic and inflammatory sequelae following a transient ischemic attack/stroke (hereby referred to collectively as 'stroke'). This study will use a powerful new technology ('hyperpolarised magnetic resonance imaging') to detect these changes in the brains of people with multiple sclerosis and Clinically Isolated Syndrome (CIS) or following a stroke when compared to a group of healthy volunteers. It will be undertaken at the University of Oxford, and each participant will undergo up to 4 scans over the course of three years.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of MS or stroke

Exclusion Criteria:

-

Max Age: 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Healthy volunteers and people with MS / stroke
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
To detect 13C metabolism in healthy participants and MS, CIS, and Stroke patients. | Baseline
  Baseline: Imaging of 13C labelled downstream metabolites from the injected metabolically active substrates in healthy participants and MS/CIS/Stroke patients, and compare to healthy volunteers

CONTACTS AND LOCATIONS:
Locations (1):
- University of Oxford, Oxford, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Upon reasonable request